CLINICAL TRIAL: NCT07114627
Title: Exploratory Study of Capecitabine Pharmacokinetics and Hand-foot Syndrome in CES1 Variant Carriers: the ESCAPE Study
Brief Title: Impact of CES1 Genotype on Capecitabine Exposure in Cancer Patients
Acronym: ESCAPE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Niels Heersche, PI: Sander Bins, Erasmus Medical Center
Other Study IDs: MEC 2024-0518; 2024-516788-96-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Solid Cancer; Gastric (Cardia, Body) Cancer; Esophageal Cancer; Colorectal Cancer (CRC)
Keywords: CAPOX; CES1; carboxylesterase 1; Capecitabine; Pharmacokinetics; Pharmacogenetics; Oncology; SNP; Single-nucleotide polymorphism; rs2244613; Hand-foot syndrome; HFS; 5-FU; ErasmusMC; Cancer
MeSH Terms: conditions — Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms; Hand-Foot Syndrome | interventions — Blood Specimen Collection; Pharmacokinetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — * Blood
  * Plasma
  * Urine
  Optional (additional consent required):
  - Skin biopt
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Single-nucleotide polymorphism (SNP): Oncological patients who are treated with CAPOX (with or without additional anti-neoplastic agents, including but not limited to nivolumab, trastuzumab or bevacizumab) according to standard of care. These patients are known carriers of the CES1 1165-33 C>A (rs2244613) SNP.
  Interventions: Drug: Blood sampling for pharmacokinetics
- Wild type: Oncological patients who are treated with CAPOX (with or without additional anti-neoplastic agents, including but not limited to nivolumab, trastuzumab or bevacizumab) according to standard of care. These patients are known carriers of the wild-type CES1 gene.
  Interventions: Drug: Blood sampling for pharmacokinetics

INTERVENTIONS:
Drug: Blood sampling for pharmacokinetics — Extra blood samples are collected for assement of the pharmacokinetics of capecitabine.

SUMMARY:
In this study, the drug capecitabine is investigated. Capecitabine is commonly used to treat breast, colon, and stomach cancers. Capecitabine is taken in tablet form. In the body, capecitabine is converted into the active molecule that has anti-cancer effects. This molecule is called 5-FU. The transformation of capecitabine to 5-FU occurs through specific proteins in the liver, also known as enzymes.

Unfortunately, capecitabine can also cause side effects. One of the most common side effects is hand-foot syndrome. In hand-foot syndrome, the palms of the hands and soles of the feet become red and painful. Previous research has shown that patients in whom one of the enzymes responsible for converting capecitabine in the liver does not function properly experience an increase in side effects frequency, particularly severe hand-foot syndrome. This specific enzyme is called CES1. It is believed that side effects occur more frequently because capecitabine is transformed more slowly, eventually leading to a prolonged exposure to 5-FU in the body.

In roughly one in three people, this enzyme functions less efficiently. To gain a better understanding of how this mechanism works, we aim to conduct this study. In this study, we will examine if patients with a less effective CES1 enzyme have higher amounts of 5-FU in their blood. We will also look into whether these patients develop side effects, such as hand-foot syndrome, more frequently. This information could eventually help us develop new strategies to reduce side effects for these patients in the future.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* 18 years of age or older;
* Planned to start treatment with concomitant capecitabine and oxaliplatin according to standard of care (irrespective of dose);
* Fit for treatment with capecitabine and oxaliplatin as judged by the treating physician;
* Capable of understanding and complying with protocol requirements and able to understand and sign the informed consent form.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Carrier of a known clinically relevant DPYD variant (i.e. *2A, *7, *13, c.1236G>A or c.2846A>T);
* Any medical condition that is known to influence capecitabine absorption (i.e. a Roux-en-Y gastric bypass operation or complete gastric resection; an esophagectomy is not considered to impair absorption);
* Prior treatment with fluoropyrimidines;
* Use of DPD-inhibitors and/or allopurinol;
* Known pregnancy at baseline.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cancer who are intended to start with CAPOX treatment.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Exposure | Up to 6 hours after intake of capecitabine
  Difference in Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC Cancer Institute, Rotterdam, Netherlands